CLINICAL TRIAL: NCT06560515
Title: Vaginal Dinoprostone Versus Vaginal Misoprostol for Induction of Labour in Post-dated Pregnancy; a Randomized Controlled Study.
Brief Title: Dinoprostone Versus Vaginal Misoprostol for Induction of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mervat Sheikhelarab Elsedeek Ibrahim Omran, Professor of Obstetrics and Gynaecology, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0107227
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Induced Vaginal Delivery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal Dinoprostone (Experimental): received 3 mg vaginal Dinoprostone of maximum 2 doses 6 hours apart.
  Interventions: Drug: Vaginal Dinoprostone
- Vaginal Misoprostol (Active Comparator): received 50μg of vaginal misoprostol of maximum 2 doses 6 hours apart.
  Interventions: Drug: Vaginal Dinoprostone

INTERVENTIONS:
Drug: Vaginal Dinoprostone — induction of labour in women with postdate pregnancy with vaginal dinoprostone vs. vaginal misoprostol

SUMMARY:
This randomized controlled study was carried out on 370 pregnant women with gestational age ≥ 40 weeks of different ages and parities at El-Shatby Maternity University Hospital after approval of ethical committee of Alexandria Faculty of Medicine. After assessment for eligibility & enrollment in the study, women were randomly assigned into one of the two study groups, Group (I) received 3 mg vaginal Dinoprostone of maximum 2 doses 6 hours apart and Group (II) received 50 μg of vaginal misoprostol of maximum 2 doses 6 hours apart.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 40 weeks or beyond
* singleton pregnancy
* Bishop score 4 or more
* fetus in a cephalic presentation
* Adequate fetal biophysical profile

Exclusion Criteria:

* Any signs of labour (Prelabor rupture of membranes)
* Grand Multiparous women (parity of 4 or more)
* IUFD
* fetal weight > 4 kg
* BMI > 35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Sucess of induction | number of women who delivered vaginally after induction
  percentage of women with a successful vaginal delivery
Induction to delivery time | time from start of induction till delivery of the fetus
  time lapse from receiving first dose of induction till delivery of the fetus

SECONDARY OUTCOMES:
Postpartum hemorrhage | after delivery of the placenta
  quantification of amount of postpartum bleeding
neonatal outcomes | at 1 and 5 minutes of delivery
  Apgar Score at 1 and 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- ElShatby University Maternal Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No